CLINICAL TRIAL: NCT06572722
Title: Perioperative Immunotherapy for Early-stage Non-small-cell Lung Cancer: a Randomised, Multicentre, Open-label, Phase 2 Trial
Brief Title: Perioperative Immunotherapy for NSCLC (ECTOP-1030)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Director in the Department of Thoracic Surgery, FUSCC, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECTOP- 1030
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — atezolizumab; Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Atezolizumab (Experimental)
  Interventions: Drug: Atezolizumab
- Nivolumab (Experimental)
  Interventions: Drug: Nivolumab
- Pembrolizumab (Experimental)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Atezolizumab — atezolizumab adjuvant therapy
  Arms: Atezolizumab
Drug: Nivolumab — nivolumab neoadjuvant therapy
  Arms: Nivolumab
Drug: Pembrolizumab — pembrolizumab neoadjuvant+adjuvant therapy
  Arms: Pembrolizumab

SUMMARY:
This trial is a randomized, multicenter, open label phase II clinical study. The main objective is to evaluate the efficacy of three perioperative immunotherapy modalities (atezolizumab adjuvant therapy, nivolumab neoadjuvant therapy, pembrolizumab neoadjuvant+adjuvant therapy) in early-stage resectable NSCLC patients. The enrolled patients are randomly assigned in a 1:1:1 ratio to receive relevant treatment in the three perioperative immunotherapy groups mentioned above, and undergoing short-term pathological efficacy evaluation and long-term prognosis follow-up after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who sign the informed consent form and are willing to complete the study according to the plan;
2. Aged from 18 to 80 years old;
3. ECOG equals 0 or 1;
4. Not receiving lung cancer surgery before;
5. Resectable cIB-IIIA tumors;
6. Not receiving chemotherapy or radiotherapy before.

Exclusion Criteria:

1. Not cIB-IIIA tumors;
2. Nodules not suitable for resection;
3. Not lung adenocarcinoma diagnosed cytologically or pathologically;
4. Receiving lung cancer surgery before;
5. Receiving radiotherapy or chemotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 2 years
  the time from randomisation to the date of first recurrence, occurrence of new primary lung cancer, or death from any cause

SECONDARY OUTCOMES:
Overall survival | 2 years
  the time from randomisation to the date of death from any cause
Major pathological response | 2 years
  ≤10% residual viable tumor cells in the primary tumor and sampled lymph nodes

CONTACTS AND LOCATIONS:
Overall Officials: Haiquan Chen, M.D., Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No